CLINICAL TRIAL: NCT02860858
Title: Intravitreal Aflibercept for Treatment of Polypoidal Choroidal Vasculopathy (PCV)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Department of Medical Services Ministry of Public Health of Thailand (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18265_CREC032/59BPs
Record Dates: First submitted 2016-07-04; First posted 2016-08-09 (Estimated); Last update posted 2020-10-23 (Actual); Status verified 2018-05

CONDITIONS: Symtomatic Macular Polypoidal Choroidal Vasculopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Aflibercept (Experimental)
  Interventions: Biological: Intravitreous aflibercept injection

INTERVENTIONS:
Biological: Intravitreous aflibercept injection

SUMMARY:
Objective: To evaluate the efficacy of intravitreal aflibercept injection on visual acuity in patients with symptomatic macular PCV.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female >/= 18 years
* Confirmed diagnosis of symptomatic macular PCV in the study eye defined by: - Active macular polypoidal lesions shown by ICGA and - Presence of serosanguinous maculopathy
* BCVA letter score between 78-24 using ETDRS visual acuity chart measured at 4 meters

Exclusion Criteria:

* Previous treatment with systemic anti-VEGF drugs within 6 months prior to Baseline (e.g., sorafenib [Nexavar®], sunitinib [Sutent®], bevacizumab [Avastin®])

Study eye:

* Active ocular inflammation or infection (ocular or periocular)
* Uncontrolled intraocular hypertension or glaucoma (IOP> 30 mmPIg) despite treatment with anti-glaucoma medication
* Predominantly-scarred PCV lesions
* Ocular disorders in the study eye (e.g. cataract, retinal vascular occlusion, diabetic retinopathy) that, in the opinion of the investigator may confound interpretation of study results or compromise VA or require medical or surgical intervention during the study period
* Prior treatment with verteporfin PDT, external-beam radiation, subfoveal or extrafoveal focal laser photocoagulation, submacular surgery, or transpupillary thermotherapy
* Prior treatment with any anti-VEGF compound or any investigational treatment
* Treatment with intravitreal or subtenon corticosteroid injection or device implantation within 90 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-12-30 (Actual); Primary Completion 2018-08-30 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Best corrected visual acuity (BCVA) | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Rajavithi Hospital, Bangkok, Thailand